CLINICAL TRIAL: NCT04700436
Title: A Multi-center, Randomized, Open-label, Active-controlled, Phase IV Clinical Trial to Evaluate the Efficacy and Safety of EzetimiBe/Rosuvastatin Diabetic Dislipidemia With Hypertriglyceridaemia
Brief Title: Efficacy and Safety of EzetimiBe/Rosuvastatin in Diabetic Dislipidemia With Hypertriglyceridaemia
Acronym: REMBRANDT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Soo Heon Kwak, Principal Investigator, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REMBRANDT
Record Dates: First submitted 2020-10-05; First posted 2021-01-07 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: Endocrine System Diseases; Nutritional and Metabolic Diseases; Diabetes Mellitus, Type 2; Dyslipidemias
MeSH Terms: conditions — Endocrine System Diseases; Nutritional and Metabolic Diseases; Diabetes Mellitus, Type 2; Dyslipidemias | interventions — Ezetimibe; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test group (Experimental): Subject administered with Rosuzet tablet 10/5 mg (Ezetimibe 10 mg/Rosuvastatin 5 mg)
  Interventions: Drug: Rosuzet tablet 10/5 mg (Ezetimibe 10 mg/Rosuvastatin 5 mg)
- Control group (Active Comparator): Subject administered with Suvast tablet 10 mg (Rosuvastatin 10 mg)
  Interventions: Drug: Suvast tablet 10 mg (Rosuvastatin 10 mg)

INTERVENTIONS:
Drug: Rosuzet tablet 10/5 mg (Ezetimibe 10 mg/Rosuvastatin 5 mg) — Test drug: Rosuzet tablet 10/5 mg (Ezetimibe 10 mg/Rosuvastatin 5 mg)
  Arms: Test group
Drug: Suvast tablet 10 mg (Rosuvastatin 10 mg) — - Control drug: Suvast tablet 10 mg (Rosuvastatin 10 mg)
  Arms: Control group

SUMMARY:
To compare and evaluate the effects of LDL-C and Triglyceride (TG) control on the first dose Ezetimibe/Statin (Rosuvastatin 5 mg/Ezetimibe 10 mg) combination therapy compared to the average dose Statin (Rosuvastatin 10 mg) monotherapy in patients with Type 2 diabetes with hypertriglyceridemia (TG > 200 mg/dL).

DETAILED DESCRIPTION:
The purpose of this study is to compare and evaluate the effects of LDL-C and Triglyceride (TG) control on the first dose Ezetimibe/Statin (Rosuvastatin 5 mg/Ezetimibe 10 mg) combination therapy compared to the average dose Statin (Rosuvastatin 10 mg) monotherapy in patients with Type 2 diabetes with hypertriglyceridemia (TG > 200 mg/dL).

ELIGIBILITY:
Inclusion Criteria:

Screening (Visit 1) Inclusion Criteria

1. Korean men and women aged 40 to 75
2. Patients who have been diagnosed with type 2 diabetes based on clinical judgment and satisfy diabetes diagnosis criteria
3. Who have the following laboratory values on an empty stomach

   * Patients with no prior statin therapy

     * Low-density lipoprotein cholesterol (LDL-C) ≥ 100 mg/dL (measured directly or calculated; calculated LDL-C is applicable only when triglyceride levels are < 400 mg/dL)
     * 200 mg/dL ≤ Triglyceride (TG) ≤ 499 mg/dL
   * Patients currently receiving low- or moderate-intensity statin therapy

     • Low-density lipoprotein cholesterol (LDL-C) ≥ 70 mg/dL (measured directly or calculated; calculated LDL-C is applicable only when triglyceride levels are < 400 mg/dL)
   * 200 mg/dL ≤ Triglyceride (TG) ≤ 499 mg/dL
4. Those with less than 9% HbA1C
5. Those who voluntarily agreed to participate in this clinical trial and signed a written ICF

Randomization (Visit 2) Inclusion Criteria

1) Persons with compliance 80% or more during Suvast tablet 5 mg Run-in period and with good TLC by investigator's judgment

Exclusion Criteria:

1. Patients with hypersensitivity to the main ingredient (Ezetimibe or Rosuvastatin) and ingredients of IP
2. Pregnant and lactating women, and women and men of childbearing potential who do not agree to conduct appropriate contraception during clinical trial
3. Patients with Body Mass Index (BMI) < 15 kg/ m2 or > 35 kg/m2
4. Persons with the following medical history or surgical/interventional history

   * Atherosclerotic disease occurring within 24 weeks at screening
   * Myopathy including rhabdomyolysis
   * Patients who have had a history of drug or alcohol abuse, or who have met drug or alcohol abuse criteria within 1 year at screening
   * Major mental illness (depression, bipolar disorder, etc.)
   * Malignant tumor within 5 years at screening
5. Persons with the following comorbidities and laboratory abnormalities

   * CK ≥ 2 X ULN
   * Patients with severe hepatopathy (AST or ALT > 5 X ULN)
   * Patients with unexplained persistent ALT elevation opinion or active liver disease
   * TSH (Thyroid stimulating hormone) > 1.5 X ULN or those who do not maintain stable thyroid stimulating hormone level by investigator's judgment
   * Uncontrolled hypertension (greater than sitBP 160/100 mmHg at screening)
   * Renal disorder patients with severe renal failure (creatinine clearance (CLcr)<30 mL/min
6. Those who have the following history of drug administration within 3 months at screening

   * Non-statin lipid modulators
   * Foods or drugs that affect lipid control
   * Systemic steroids
7. Those who are expected to administer contraindication drugs during clinical trial, including screening
8. Those who have persistent history of drinking within 1 week at clinical trial participation or who are unable to perform TLC due to continuous drinking during clinical trial
9. Patients with genetic problems such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorptioin
10. Those who received other IPs or investigational medical devices within 30 days at screening
11. Patients judged to be ineligible to participate in clinical trial by investigator's decision

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2020-01-03 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2024-02-13 (Actual)

PRIMARY OUTCOMES:
LDL-C change rate (percent, %) | Baseline and 16 weeks
  To compare LDL-C change rate (percent, %) between test and control group
Triglyceride (TG) change rate (percent, %) | Baseline and 16 weeks
  To compare Triglyceride (TG) change rate (percent,%)between test and control group

SECONDARY OUTCOMES:
Change rates (percent, %) of LDL-C and Triglyceride (TG) | Baseline and 4 weeks
  To measure/compare Change rates (percent, %) of LDL-C and Triglyceride (TG) between test and control group
Changes (mg/dL) of Total cholesterol (TC), Triglyceride (TG), HDL-C, and non-HDL-C | Baseline, 4 weeks, and 16 weeks
  To measure/compare Changes (mg/dL) of Total cholesterol (TC), Triglyceride (TG), HDL-C, and non-HDL-C between test and control group
Percent (%) of subjects with a 50% or more reduction in LDL-C level | 4 weeks and 16 weeks
  To measure/compare Percent (%) of subjects with a 50% or more reduction in LDL-C level between test and control group
Percent (%) of subjects with LDL-C below 70 mg/dL | 4 weeks and 16 weeks
  To measure/compare Percent (%) of subjects with LDL-C below 70 mg/dL between test and control group
Changes of lipoproteins (ApoA1, ApoB) | Baseline and 16 weeks
  To measure/compare Changes of lipoproteins (ApoA1 (mg/dL), ApoB (mg/dL)) between test and control group
Changes of lipoproteins (ApoB/ApoA1 ratio) | Baseline and 16 weeks
  To measure/compare Changes of lipoproteins (ApoB/ApoA1 ratio) between test and control group
Change of HOMA-IR | Baseline and 16 weeks
  To measure/compare Change of HOMA-IR between test and control group
Change of HbA1C (percentage, %) | Baseline, 4 weeks, and 16 weeks
  To measure/compare Change of HbA1C (percentage, %) between test and control group
Change (mg/dL) of Fasting Plasma Glucose (FPG) | Baseline, 4 weeks, and 16 weeks
  To measure/compare Change (mg/dL) of Fasting Plasma Glucose (FPG) between test and control group
Change (mg/dL) of hs-CRP | Baseline and 16 weeks
  To measure/compare Change (mg/dL) of hs-CRP between test and control group
Changes of plasma triglyceride (mg/dL), ApoB100 (mg/dL), and ApoB48 (mg/dL) levels at 30-minute, 1-, 2-, 3-, 4-, 5-, and 6-hour before and after FMC in subjects who perform FMC | Baseline and 16 weeks
  To measure/compare Changes of plasma triglyceride (mg/dL), ApoB100 (mg/dL), and ApoB48 (mg/dL) levels at 30-minute, 1-, 2-, 3-, 4-, 5-, and 6-hour before and after FMC in subjects who perform FMC between test and control group
On the graphs at 30-minute, 1-, 2-, 3-, 4-, 5-, and 6-hour before and after FMC in subjects who perform FMC, total Area Under the Curve (tAUC) of each plasma triglyceride (mg/dL), ApoB100 (mg/dL), and ApoB48 (mg/dL) | Baseline and 16 weeks
  To measure/compare On the graphs at 30-minute, 1-, 2-, 3-, 4-, 5-, and 6-hour before and after FMC in subjects who perform FMC, total Area Under the Curve (tAUC) of each plasma triglyceride (mg/dL), ApoB100 (mg/dL), and ApoB48 (mg/dL) between test and control group
Adverse event | Baseline and 16 weeks
  To measure/compare Adverse event between test and control group
Blood pressure | Baseline and 16 weeks
  To measure/compare Blood pressure between test and control group
Pulse | Baseline and 16 weeks
  To measure/compare Pulse between test and control group
Electrocardiogram (12-lead ECG) | -4 weeks and 16 weeks
  Number(%) of participants with Clinically Significant or Normal Electrocardiogram (12-lead ECG) findings after study drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Kyong Soo Park, Dr., Principal Investigator — Principal Investigator
Locations (26):
- South Korea (26):
  - Korea University Ansan Hospital, Ansan
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si
  - Soon Chun Hyang University Hospital Cheonan, Cheonan
  - Keimyung University Dongsan Medical Center, Daegu
  - Yeongnam University Medical Center, Daegu
  - Eulji University Hospital, Daejeon
  - Kyung Hee University Hosipital at Gangdong, Gangdong
  - Inje University Ilsan Paik Hospital, Goyang-si
  - Hanyang University Guri Hospital, Guri-si
  - Chosun University Hospital, Gwangju
  - Hallym University Medical Center-Dongtan, Hwaseong-si
  - Inha University Hospital, Inchon
  - Pusan National University Hospital, Pusan
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Kyung Hee University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - The Catholic University of Korea, Seoul St.Mary, Seoul
  - The Catholic University of Korea, Yeouido St. Mary's Hospital, Seoul
  - Yonsei University Health System, Gangnam Severance Hospital, Seoul
  - Yonsei University Health System, Severance Hospital, Seoul
  - Gachon University, Donginchoen Gil Hospital, Sŏngnam
  - Seoul National University Bundang Hospital, Sŏngnam
  - Ajou University Hospital, Suwon
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon

IPD SHARING:
Plan to Share IPD: No